CLINICAL TRIAL: NCT02765399
Title: The Effect of Liraglutide Treatment on Postprandial Chylomicron and VLDL Kinetics, Liver Fat and de Novo Lipogenesis - a Single-center Randomized Controlled Study
Brief Title: The Effect of Liraglutide Treatment on Postprandial Chylomicron and VLDL Kinetics, Liver Fat and de Novo Lipogenesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Niina Matikainen, Senior Endocrinologist, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIRA
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Liraglutide (Experimental): Liraglutide subcutaneous injection once daily with following dose escalation:
  liraglutide 0.6 mg once daily for one week; liraglutide 1.2 mg once daily for one week and thereafter liraglutide 1.8 mg once daily for 3.5 months.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo subcutaneous injection once daily with following dose escalation:
  placebo 0.1 ml once daily for one week; placebo 0.2 ml once daily for one week and thereafter placebo 0.3 ml once daily for 3.5 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study aims to evaluate the mechanisms underlying the effect of incretin therapy on lipoprotein metabolism in subjects with type 2 diabetes and to study the effect of liraglutide on hepatic de novo lipogenesis.

DETAILED DESCRIPTION:
The well recognized dyslipidemia in people with type 2 diabetes consists of high fasting and non-fasting plasma triglycerides (TG), low high-density lipoprotein (HDL) -cholesterol and preponderance of small dense low-density lipoprotein (LDL) particles nominated as the atherogenic lipid triad. Humans are mostly in a postprandial rather than fasting state and therefore non-fasting TG values reflect more accurately the continuous exposure of arterial wall to triglyceride rich lipoproteins (TRLs) and more importantly, to substantial cholesterol load that these particles deliver.

Postprandial lipemia is highly prevalent even in type 2 diabetes patients with normal fasting TG concentrations. Intestinal overproduction of chylomicrons (CMs) and the structural protein apolipoprotein (apo)-B48 has been identified as an integral feature of postprandial lipemia in type 2 diabetes and insulin resistance. It is clinically important to elucidate the mechanism for delayed postprandial lipemia and the interactions between dysglycemia and dyslipidemia in type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes treated with a lifestyle or metformin (any dose)
* waist circumference > 88 cm in women and > 92 cm in men
* BMI 27-40 kg/m2
* triglycerides between 1.0 - 4.0 mmol/L
* LDL < 4.5 mmol/l

Exclusion Criteria:

* Type 1 diabetes
* Apo E2/2 phenotype
* ALT/AST > 3x ULN
* GFR < 60 ml/min, clinically significant TSH outside normal range
* Lipid-lowering drugs other than statins within 6 months
* Current treatment with pioglitazone, insulin, sulphonylureas, gliptins, glinides, SGLT-2 inhibitors or thiazide diuretics (at a dose of > 25 mg / day)
* Blood pressure > 160 mmHg systolic and/or > 105 diastolic
* History of pancreatitis or stomach / other major bleeding, thyroid neoplasia, persistent hypothyroidism or persistent hyperthyroidism
* Any medical condition that puts the patient in the risk of dehydration
* Concurrent medical condition that may interfere with the interpretation of efficacy and safety data during the study.
* Females of childbearing potential who are not using adequate contraceptive methods
* Subjects who have experienced side-effects previously from GLP-1 agonists
* Non-compliance or withdrawal of consent
* Any information or clinical event described in liraglutide SPC that is a contraindication for the use of liraglutide

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niina Matikainen, MD, PhD, Principal Investigator — Senior Endocrinologist
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zech LA, Grundy SM, Steinberg D, Berman M. Kinetic model for production and metabolism of very low density lipoprotein triglycerides. Evidence for a slow production pathway and results for normolipidemic subjects. J Clin Invest. 1979 Jun;63(6):1262-73. doi: 10.1172/JCI109421. PMID 221537
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] Kernan WN, Inzucchi SE, Viscoli CM, Brass LM, Bravata DM, Shulman GI, McVeety JC, Horwitz RI. Pioglitazone improves insulin sensitivity among nondiabetic patients with a recent transient ischemic attack or ischemic stroke. Stroke. 2003 Jun;34(6):1431-6. doi: 10.1161/01.STR.0000071108.00234.0E. Epub 2003 May 1. PMID 12730556
- [Result] Matikainen N, Soderlund S, Bjornson E, Pietilainen K, Hakkarainen A, Lundbom N, Taskinen MR, Boren J. Liraglutide treatment improves postprandial lipid metabolism and cardiometabolic risk factors in humans with adequately controlled type 2 diabetes: A single-centre randomized controlled study. Diabetes Obes Metab. 2019 Jan;21(1):84-94. doi: 10.1111/dom.13487. Epub 2018 Sep 4. PMID 30073766
- [Result] Taskinen MR, Bjornson E, Matikainen N, Soderlund S, Pietilainen KH, Ainola M, Hakkarainen A, Lundbom N, Fuchs J, Thorsell A, Andersson L, Adiels M, Packard CJ, Boren J. Effects of liraglutide on the metabolism of triglyceride-rich lipoproteins in type 2 diabetes. Diabetes Obes Metab. 2021 May;23(5):1191-1201. doi: 10.1111/dom.14328. Epub 2021 Mar 5. PMID 33502078
- [Result] Bjornson E, Packard CJ, Adiels M, Andersson L, Matikainen N, Soderlund S, Kahri J, Sihlbom C, Thorsell A, Zhou H, Taskinen MR, Boren J. Investigation of human apoB48 metabolism using a new, integrated non-steady-state model of apoB48 and apoB100 kinetics. J Intern Med. 2019 May;285(5):562-577. doi: 10.1111/joim.12877. Epub 2019 Mar 12. PMID 30779243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 54 subjects were assessed for eligibility, of whom 31 were excluded because of failure to meet inclusion criteria (n = 28) or declining to participate (n = 1), or for other reasons (n = 2).
Groups:
- Liraglutide: Liraglutide subcutaneous injection once daily with following dose escalation:
  liraglutide 0.6 mg once daily for one week; liraglutide 1.2 mg once daily for one week and thereafter liraglutide 1.8 mg once daily for 3.5 months.
  Liraglutide
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 16 | 7
Completed | 15 | 7
Not Completed | 1 | 0
Not completed — Nausea | 1 | 0

BASELINE CHARACTERISTICS:
Population: In total, 54 subjects were assessed for eligibility, of whom 31 were excluded because of failure to meet inclusion criteria (n=28) or declining to participate (n=1), or for other reasons (n=2). In total, 22 participants completed the first study. One participant in the liraglutide arm discontinued the study at Week 7 because of nausea. None of the other participants reported adverse effects during the study, with the exception of mild nausea.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 16 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 7 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 14 | 3 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 7 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Finland | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Liver Fat Content
Description: Before vs after intervention (Liraglutide or placebo): mean liver fat content was measured by magnetic resonance imaging. Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: fat %
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
fat %
  Baseline | 14.8 (7.4) | 16.1 (9.3)
  16 weeks | 10.7 (6.3) | 13.9 (9.7)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.028, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Plasma Triglyceride (TG) Area Under Curve (AUC)
Description: Before vs after intervention (Liraglutide or placebo): postprandial plasma TG summary measured using the trapezoidal rule and expressed as AUC (at fasting and at 0.5, 1, 2, 3, 4, 6 and 8 hours) after oral fat tolerance test. Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: mmol/l per h
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
mmol/l per h
  Baseline | 22.0 (7.4) | 17.5 (4.8)
  16 weeks | 17.1 (5.0) | 19.0 (6.2)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.011, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.612, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Body Weight
Description: Before vs after intervention (Liraglutide or placebo): Change in body weight. Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
kg
  Baseline | 98.6 (11.0) | 92.0 (7.4)
  16 weeks | 96.1 (11.2) | 89.8 (6.3)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.128, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in HbA1c Level
Description: Before vs after intervention (Liraglutide or placebo): Change in B -Hemoglobiini-A1c level in plasma. Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: HbA1c %
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
HbA1c %
  Baseline | 7.0 (1.0) | 6.3 (0.3)
  16 weeks | 6.4 (0.7) | 6.4 (0.5)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.343, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Change in fP-glucose Level
Description: Before vs after intervention (Liraglutide or placebo): concentration of fasting plasma glucose measured using the hexokinase method. Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
mmol/L
  Baseline | 8.3 (2.4) | 6.5 (0.8)
  16 weeks | 6.4 (1.2) | 6.4 (0.9)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.865, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Change in Insulin Level
Description: Before vs after intervention (Liraglutide or placebo): Concentration of insulin level in plasma measured using electrochemiluminescence. Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after16 weeks
Measure: Mean (Standard Deviation); unit: μU/mL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
μU/mL
  Baseline | 13.9 (4.8) | 13.8 (6.9)
  16 weeks | 14.5 (4.9) | 14.1 (5.5)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.532, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.735, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Change in Matsuda Index
Description: Before vs after intervention (Liraglutide or placebo): Matsuda index was calculated for assessment of insulin sensitivity in plasma at time points 0, 30, 60 and 120 minutes using formula 10,000/square root of [fasting glucose x fasting insulin] x [mean glucose x mean insulin during oral glucose tolerance test]. The Matsuda index is considered to be the gold standard to determine insulin sensitivity without glucose clamp studies (Matsuda M, DeFronzo RA. Diabetes Care. 22:1462-70). Subjects who don't have insulin resistance have values of Matsuda Index of 2.5 or higher (Kerman WN et al. Stroke 34:1431;2003). Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
index
  Baseline | 2.5 (1.0) | 3.1 (1.7)
  16 weeks | 3.5 (1.8) | 3.1 (1.3)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.753, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Change in VAT Area
Description: Before vs after intervention (Liraglutide or placebo): visceral adipose tissue area measured by magnetic resonance imaging (MRI). Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
cm3
  Baseline | 3403 (941) | 2710 (836)
  16 weeks | 3185 (1014) | 2600 (825)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.047, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.499, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Change in SAT Area
Description: Before vs after intervention (Liraglutide or placebo): subcutaneous adipose tissue area measured by magnetic resonance imaging (MRI). Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
cm3
  Baseline | 4043 (1129) | 5400 (1598)
  16 weeks | 3792 (1185) | 5161 (1653)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.128, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Change in ApoCIII Level
Description: Before vs after intervention (Liraglutide or placebo): apolipoprotein CIII concentration in plasma measured by using turbidimetric immunoassay. Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
mg/dL
  Baseline | 12.0 (4.4) | 9.7 (2.8)
  16 weeks | 9.9 (3.7) | 8.6 (1.8)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.018, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.578, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Hepatic de Novo Lipogenesis
Description: Before vs after intervention (Liraglutide or placebo): Hepatic DNL is calculated from enrichment of deuterated water ingested during the kinetic study at specified time points (0, 4 and 8 hrs.). Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
μmol/L
  Baseline | 15.4 (7.4) | 12.6 (7.5)
  16 weeks | 19.1 (13.1) | 13.8 (11.2)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.152, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.866, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in Systolic RR
Description: Before vs after intervention (Liraglutide or placebo): systolic blood pressure measurements. Results from Matikainen et al. Diabetes Obes Metab 21:84-94; 2019.
Time Frame: Baseline and after 16 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 7
mm Hg
  Baseline | 135 (14) | 145 (10)
  16 weeks | 139 (11) | 137 (11)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.173, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.018, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Mean Total Production of apoB48
Description: Before vs after intervention (Liraglutide or placebo): ApoB48 total production in plasma measured by using multicompartmental modeling. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (JCI 63:1262;1979) and have been widely used over 30yrs. So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. JIM 285:562;2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al. Diabetes Obes Metab. 23:1191; 2021.
Time Frame: Baseline and after 16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
mg/day
  Baseline | 490 (190) | 570 (68)
  16 weeks | 329 (140) | 530 (120)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 1, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Mean Production Rate of apoB48 in CM
Description: Before vs after intervention (Liraglutide or placebo): Change in mean production rate of ApoB48 in chylomicrons isolated from plasma samples and measured by multicompartmental modeling assay. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (JCI 1979). So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. JIM 2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al.
Time Frame: Baseline and after 16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
mg/day
  Baseline | 284 (130) | 190 (35)
  16 weeks | 113 (53) | 160 (57)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.79, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Mean apoB48 FTR to VLDL1 Particles
Description: Before vs after intervention (Liraglutide or placebo): Change in apoB48 chylomicron fractional transfer rate to VLDL1 isolated from plasma by ultracentrifugation and by liquid chromatography/mass spectrometry and calculated with multicompartmental modeling assay. So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. JIM 2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al. 2021.
Time Frame: Baseline and after 16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: pools/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
pools/day
  Baseline | 12 (4) | 34 (12)
  16 weeks | 26 (13) | 30 (10)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.13, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Mean TG Fractional Catabolic Rates in CM
Description: Before vs after intervention (Liraglutide or placebo): Change in triglycerides fractional catabolic rates in isolated chylomicrons from plasma samples measured by multicompartmental modeling assay. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (JCI 1979). So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. JIM 2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al. DOM 2021.
Time Frame: Baseline and after 16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: pools/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
pools/day
  Baseline | 33 (13) | 64 (15)
  16 weeks | 46 (20) | 59 (12)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.011, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.13, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Mean CM FDC of apoB48
Description: Before vs after intervention (Liraglutide or placebo): Change in chylomicron fractional direct clearance rates of apoB48 measured from plasma by liquid chromatography - mass spectrometry with multicompartmental modeling assay. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (1979). So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. 2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al. 2021.
Time Frame: Baseline and after 16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: pools/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
pools/day
  Baseline | 9 (5) | 4.4 (1.6)
  16 weeks | 0.8 (0.4) | 3.2 (2.5)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.13, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Change in Direct CM-apoB48 Clearance
Description: Before vs after intervention (Liraglutide or placebo): Direct apoB48 clearance rates in isolated chylomicrons and measured by liquid chromatography - mass spectrometry and calculated by multicompartmental modeling assay. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (1979). So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. 2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al. 2021.
Time Frame: Baseline and after 16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
mg/day
  Baseline | 106 (63) | 20 (3.8)
  16 weeks | 3.8 (2.5) | 17 (12)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.79, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Mean CM-apoB48 Transfer Rates to VLDL1
Description: Before vs after intervention (Liraglutide or placebo): Change in chylomicron-apoB48 transfer rates to VLDL1 isolated from plasma by ultracentrifugation and measured using multicompartmental modeling. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (1979). So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. 2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al. 2021.
Time Frame: Baseline and after 16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
mg/day
  Baseline | 127 (120) | 170 (38)
  16 weeks | 110 (57) | 150 (50)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.79, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Mean VLDL1-TG Production Rates
Description: Before vs after intervention (Liraglutide or placebo): Change in VLDL1 production rates measured from isolated VLDL from plasma samples by ultracentrifugation and measured using mathematical modeling. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (JCI 1979). So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. JIM 2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al. DOM 2021.
Time Frame: Baseline and after16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
g/day
  Baseline | 51 (21) | 43 (1.7)
  16 weeks | 35 (9.8) | 35 (10)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.18, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Mean Fractional Catabolic Rate of VLDL2-apoB100
Description: Before vs after intervention (Liraglutide or placebo): Change in VLDL2-apoB100 fractional catabolic rates measured from isolated VLDL2 from plasma by ultracentrifugation and measured using mathematical modeling. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (JCI 1979). So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. JIM 2019). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90,120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. Results from Taskinen et al. DOM 2021.
Time Frame: Baseline and after 16 weeks
Population: 18 subjects only volunteered to the kinetic study.
Measure: Mean (Standard Deviation); unit: pools/day
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 14 | 4
pools/day
  Baseline | 6.7 (2.6) | 4.5 (2)
  16 weeks | 5.6 (2.2) | 5.1 (2.1)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Other; p = 0.068, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.63, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During 16 weeks of Liraglutide therapy
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/7
Other Adverse Events (participants affected / at risk) | 4/16 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liraglutide (N=16) | Placebo (N=7)
Nausea (General disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT02765399/Prot_SAP_000.pdf